CLINICAL TRIAL: NCT04764487
Title: A Web-mediated Follow-up With the Web-application KidneyPRO Versus Standard Follow-up for Patients With Advanced Renal Cell Carcinoma Treated With Axitinib/Pembrolizumab in First Line
Acronym: AxiPRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Collaborators: Pfizer (Industry); FLGXPL (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WP-2019-03; 2020-A01103-36 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Renal Cell Carcinoma Metastatic
Keywords: Web-application; Quality Of Life; Metastatic renal cell carcinoma; Follow-up; Progression Free Survival; Overall Survival
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard follow-up (Other): Patients will have no intervention. It is the comparator group. Patients will have the usual follow-up for clinical, biological and imaging exams.
  Interventions: Other: standard follow-up
- KidneyPRO web-application follow up (Experimental): Patients will have to connect to the KidneyPRO web-application weekly to complete a questionnaire about their symptoms in addition to usual follow-up.
  Appropriate care will be offered if necessary (depending on the symptoms assessment)
  Interventions: Device: KidneyPRO

INTERVENTIONS:
Device: KidneyPRO — Web-application for symptoms assessment
  Other Names: web-application
  Arms: KidneyPRO web-application follow up
Other: standard follow-up — usual follow-up
  Arms: Standard follow-up

SUMMARY:
With the advent of immunotherapy, standard first-line treatment for patients with renal cell carcinoma is now an association with an immune checkpoint inhibitor. In this context, the association axitinib plus pembrolizumab has already been evaluated in several studies with positive results for Progression Free survival, Overall survival and Complete response. The combo received a positive opinion from the Committee for Medicinal Products for Human Use, and the European Commission approves the extension of Marketing Authorization in first line for metastatic renal cell carcinoma patients.

In a context of treatment with a new association, it is important to manage the toxicities closely in order to allow the patients to have an optimal treatment. The underlying hypothesis is that the use of new information and communication technologies could improve clinical patient management.

In this study, we wish assess the impact of monitoring via the web application KidneyPRO on the quality of life of patients with the new combination of treatment axitinib/pembrolizumab for a renal cell carcinoma in first line.

DETAILED DESCRIPTION:
Metastatic or locally advanced clear cell renal carcinomas (RCC) are treated with targeted therapies (inhibitors of tyrosine kinases) and immune check-points inhibitors.

In first line many combos are tested. Association of TKI-PD L1-inhibitor is one option. Axitinib-Pembrolizumab showed very high response rate and progression free survival compared to Sunitinib but immunotherapies have a specific adverse event profile. Actually, there is no standardized follow-up for this type of treatment.

It is important to develop new strategies that reduce the resources used while improving the performance of this surveillance for the benefit of patients, to improve the comfort of patients, to improve the compliance and to optimise the dose of treatment received, in a course of care reworked by maintaining a continuous contact not demanding.

In collaboration with the Scientific Research National Center, the theory of chaos and its derivatives was applied to cancer and a web-application was developed on these concepts to remotely analyze the dynamics of the symptoms felt by the patient and early detect a recurrence or a complication of his cancer. Clinical symptoms are self-assessed by patients once a week, transcribed on their smartphone or computer through the Internet application. Relevant clinical events are detected using data processing algorithms, combining the dynamics of the various reported symptoms. In this case, an alert message is sent to the health care team. The referring oncologist is thus warned early. He can then make a telephone call to the patient about the reality of the medical alert and summon him for a check-up or any other complementary examination.

Applied to lung cancer, this application is a tried-and-tested solution with a phase III clinical trial. The main criteria was overall survival. The monitoring of these patients with the web-application and with a number of scanners reduced by 50% compared to the reference arm, made it possible to diagnose relapses earlier, to treat them under better conditions and, above all, to improve statistically significant overall survival (a gain in overall survival of 26% at 1 year (in patients intending to treat): 49% in the standard arm versus 75% in the experimental arm: p = 0.0025. This profit persists with 2 years of decline (a median gain in overall survival of 7.6 months, p=0.0312).

This concept was confirmed in the NCT0578006 study published by Basch et al. Basch used a similar application during chemotherapy treatment in 766 cancer patients. The web-application has improved overall survival by 5 months (Hazard ratio: 0.83).

This web-application provided a statistical improvement in the quality of life for lung cancer, access to new therapeutic lines (74% versus 33%, p <0.001) and optimally with treatments delivered at therapeutic doses (in 76% versus 34%) and faster access to supportive care for a clear improvement in the general condition of patients (77 versus 33%, p <0.001). The key for these patients who experienced many treatment toxicities was to use a better method of active follow-up.

A real-time survey of quality of life of Renal Cell Cancer patients receiving Axitinib/Pembrolizumab is an objective that has never been evaluated. This study will allow to generate data in patients who were not included in the phase III study (KEYNOTE 426): Performance Status =2, with central nervous system metastasis and with renal insufficiency. Personalized monitoring of these patients with the web-application KidneyPRO is even more relevant because the aim would be to quickly provide care adapted to adverse events, supportive care in case of loss of activity…

The web-application KidneyPRO investigated has been developed for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced RCC who require a first line systemic treatment by axitinib/pembrolizumab combo
2. Patient with at least one measurable lesion according to RECIST 1.1 criteria or with clinically apparent disease that can be reliably monitored by the investigator
3. Patient aged 18 years or older
4. Eastern Cooperative Oncology Group (ECOG) Performance Status < 3
5. Patient with adequate hematopoietic or organ function, as indicated by the following criteria (assessed within -14 days prior the first dosing):

   * WBC > 2 x 109/L
   * Polynuclear neutrophils > 1.5 x 109/L
   * Platelets > 100 x 109/L
   * Hemoglobin > 8.0 g/mL
   * ALT/AST < 2.5 x ULN in the absence of liver metastases or < 5x ULN in the presence of liver metastases
   * Bilirubin < 1.5 x ULN (except Gilbert Syndrome: < 3.0 mg/dL)
   * Creatinine clearance ≥ 30 mL/min (measured or calculated by Cockroft and Gault formula) or serum creatinine < 2.0 x ULN
6. Patient possessing an initial symptom score less than or equal to 6 (Specific scale: assessment of the importance of 3 symptoms in appendix 1)
7. Patient has internet access and an email account (or has someone at home who can help send patients' symptoms or complete the form)
8. Woman of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the first administration of study treatment.
9. Patients who are sexually active must agree to use a highly effective method of contraception (e.g. implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner, for participating women; condoms for participating men) or practice complete abstinence, beginning 14 days before the first administration of study treatment, while on treatment.
10. Patient without symptomatic brain metastases (non-symptomatic metastases : without edema, not on corticosteroids, not eligible for radiation therapy/surgery and not receiving active treatments).
11. Patient enrolled in social security
12. Patient has given his written consent ahead of any specific protocol procedure

Exclusion Criteria:

1. Prior systemic therapy directed at advanced or metastatic RCC
2. Patient with contraindication to a treatment by axitinib/pembrolizumab
3. Prior immunotherapy with IL-2, IFN-α, or anti PD 1, anti PD L1, anti PD L2, anti CD137 or anti cytotoxic T lymphocyte associated antigen 4 (CTLA 4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T cell co stimulation or immune checkpoint pathways or TKI
4. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partially controlled asthma Global Initiative for Asthma 2011)
5. Uncontrolled hypertension in spite of anti-hypertensive therapy
6. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
7. Any of the following in the previous 6 months: deep vein thrombosis or symptomatic pulmonary embolism
8. Current use of immunosuppressive medication, EXCEPT for the following:

   1. intranasal inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
   2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered as a form of systemic treatment
10. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo/hyperthyroid diseases not requiring immunosuppressive treatment are eligible
11. Prior organ transplantation including allogenic stem-cell transplantation
12. Active serious infections requiring systemic antibiotic or antimicrobial therapy
13. Known history of testing positive for HIV or known acquired immunodeficiency syndrome
14. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
15. History of pneumonitis that required steroids, or current pneumonitis
16. Vaccination within 4 weeks of the first dose of pembrolizumab and while on trial is prohibited except for administration of inactivated vaccines (for example, inactivated influenza vaccines)
17. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis
18. Patient deprived of their liberty, under guardianship or trusteeship
19. Patient is being treated for another cancer and has not been cured
20. Patient with dementia, mental disorders or psychological pathology which could compromise patient informed consent and/or the observance of the study protocol
21. Patient cannot submit to the protocol for psychological, social, familial or geographical reasons
22. Patient is pregnant or breastfeeding
23. Patient is participating in another interventional study of telemonitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-06-07 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
symtom specific Quality Of Life at 24 weeks | 6 months
  difference of 4 points of the Quality Of Life, between the two arms, by the FACT-Kidney Symptom Index (FKSI-19) 24 weeks (6 months) after the first treatment administration date. Higher score is worse.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Calculated from the date of randomization to the date of death due to any cause or the date last known to be alive if patient is censored.
Progression Free survival | 2 years
  Calculated from the date of start of treatment to the date of first progression of disease based on Investigator assessment or the date of death or censored at the date of the last valid tumor assessment before start of a new therapy for patients who are still alive and without progression
Treatment Free Survival | 2 years
  Evaluated from the date of last administration of treatment to the date of the first administration of the next line of treatment or the date last known to be alive if patient is censored
Duration Of Response | 2 years
  Evaluated from the date of the first documented tumor response to the date of disease progression or the date last known to be alive if patient is censored
Change From Baseline in FACT-Kidney Symptom Index (FKSI)-19 | 2 years
  TThe FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains- Disease Related Symptoms (physical and emotional), Treatment related side effects and Functional and Well-Being . A negative change from Baseline represents a worsening of condition.
Change From Baseline in Quality Of life Questionnaire-C30 (QLQ-C30) | 2 years
  QLQ-C30 is a generic questionnaire for cancer patients. Score will be calculated according to European Organisation for Research and Treatment of Cancer guidelines for QLQ-C30. . QoL with QLQ-C30 will be evaluated before start of treatment and every 3 months until 24 months and at the end of treatment. A negative change from Baseline represents a worsening of condition.
Number of patients who experienced an adverse event (AE) | 2 years
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Duration of the treatment | 2 years
  Calculated from the date of the first administration of the treatment until the last administration of the last treatment in progress
Time to treatment discontinuation/failure due to toxicity | 2 years
  Calculated from the date of the first administration of the treatment until the date of the first discontinuation / failure due to toxicity of one of the 2 molecules
Description of subsequent cancer treatments | 2 years
  Names of subsequant cancer treatments
Web-application compliance | 2 years
  evaluated by the following ratio: the number of completed questionnaires made via the app verus the theoretical number of questionnaires that the included patients should have complete during a given period
Treatment compliance | 2 years
  Evaluated by the number of taken tablets verus.the theoretical number of tablets the patient should have taken during a given period
Sensibility of the application | 2 years
  Evaluated the number of events diagnosed by the app on the number of events that occurred in total.
Patient web-application satisfaction | 1 year
  Evaluated by a specific self-evaluation at the 6th and 12th month follow-up visits (specific questionnaire dedicated to the use of the web-application) and at the end of treatment
Performance Status at the end of treatment | 2 years
  Evaluated with the Eastern Cooperative Oncology Group's recommendations, at each visit
Medical team web-application satisfaction | 1 year
  Evaluated with a specific questionnaire at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Eric VOOG, MD, Principal Investigator — Clinique Victor Hugo/Centre Jean Bernard
Locations (13):
- France (13):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU Jean Minjoz, Besançon
  - Clilnique Pasteur, Brest
  - CHRU Brest, Brest
  - Centre François Baclesse, Caen
  - CHD Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo / Centre Jean Bernard, Le Mans
  - Centre Léon Bérard, Lyon
  - Institut Jean Godinot, Reims
  - CHP St Grégoire, Saint-Grégoire
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No